CLINICAL TRIAL: NCT07305701
Title: Mental Health of Medical Students in Orleans: a Cohort Study of a New Faculty
Brief Title: Cohort Study on Medical Students' Mental Health
Acronym: OSMOSE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHUO-2025-10
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder; Suicidal Ideation; Alcoholism; Marijuana Abuse; Loneliness
Keywords: Students; Medical students; depression; epidemiology
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Suicidal Ideation; Alcoholism; Marijuana Abuse; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical students: Medical students: students who succeed to integrate medical school after the selection at the end of the first year of health studies.
  Interventions: Other: Questionnaire
- Non medical students: Non medical students: students who fail to integrate medical school after the selection at the end of the first year of health studies.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire to be completed once a year

SUMMARY:
The main objective of this study is to identify risk factors for depression among medical students by comparing them to students who completed their first year but did not enter the medical program (students not accepted into the second year of medical school).

Major Depressive Disorder (MDD) will be assessed using a validated tool: the Composite International Diagnostic Interview Short-Form (CIDI-SF).

This a prospective, longitudinal, cohort study. The plan is to inform each new cohort of students at the Orléans University Hospital medical school for 10 years. It is estimated that 5,000 to 10,000 students will be able to participate in the study.

A link to access the study questionnaire will be sent to students by email via the registrar's office, with one email per week for four weeks. The email will contain a link to a web page where the questionnaire can be completed. The questionnaire will be available online on computers or smartphones for six weeks: from mid-October to the end of November. The questionnaire will be completed each year for the duration of the study or until the student completes their studies.

Duration of the inclusion period: 10 years Duration of participation for each participant: maximum 12 years Total duration of the study: 22 years As the cohort progresses, longitudinal analyses may be conducted to study the evolution of various disorders over time, adjusting for known confounding factors. Following the initial analyses of this study, a new interventional study will be set up to identify students at risk and offer them appropriate care.

DETAILED DESCRIPTION:
The COVID-19 pandemic has led to an increase in depression, particularly among younger people. The French Health Barometer, conducted every 4-5 years by Santé Publique France (SPF), found that the prevalence of a major depressive disorder (MDD) among 18-25 years old doubled (from 11.7% to 20.8%) between 2017 and 2021. There has also been an increase in suicidal thoughts and suicide attempts. Among students, data from the 2016 of observatoire de la vie étudiante (OVE) showed a higher prevalence of MDD and suicidal thoughts among students compared to the general population of the same age group. For medical students, a national study conducted in 2021 revealed rates of depression and suicidal thoughts far exceeding those of the general population of the same age. Financial difficulties were the main factor associated with the risk of depression. Indeed, students are a particularly vulnerable population to precariousness due to several factors. Economically, they often have limited income, relying on parental support, insufficient scholarships, or precarious jobs. This exposes them to difficulties in meeting essential needs such as housing, food, and healthcare. Socially, isolation can worsen their situation, especially when they move away from their family network or faced with academic pressure. Furthermore, high academic demands combined with unstable living conditions affect their mental health and may contribute to the development of psychiatric disorders, often untreated due to lack of resources or accessible care. This multidimensional precariousness highlights the need for comprehensive support for this population, especially since students rarely seek professional help. In the 2021 survey, only 32% of medical students suffering from depression received adequate care. To improve the health of medical students, it is therefore not enough to treat disorders; we must also prevent their onset by helping students achieve a state of well-being.

This a prospective, longitudinal, cohort study aims is to identify risk factors for depression among medical students by comparing them to students who completed their first year but did not enter in the medical program (students not accepted into the second year of medical school). The main objective of this study is to assess Major Depressive Disorder (MDD) using a validated tool : the Composite International Diagnostic Interview Short-Form (CIDI-SF).

We will assess the 12-month prevalence of the main psychiatric disorders evaluated, dropout using a single question, and loneliness. Care utilization will be measured, as well as care avoidance and its causes, along with financial and social insecurity, educational satisfaction, and stigma. Additional variables or questionnaires may be added through protocol amendments. These measurements will be obtained through students filling out an online questionnaire. Quantitative analyses will be conducted, starting with univariate and then multivariate models, with adjustments for known confounding factors.

The plan is to inform each cohort of students at the Orléans University Hospital medical school for 10 years. It is estimated that 5,000 to 10,000 students will be able to participate in the study.

Each year, all medical students will be informed of the protocol at meetings at the University of Orléans at the start of the academic year in September regardless of their year of study (e.g. 1st year of medical study, 2nd, 3rd, 4th year of study etc…). The study will be offered each year to students entering PASS/LAS at the Faculty of Medicine of the University of Orléans and to cohorts that have already begun their medical studies.

A link to access the study questionnaire will be sent to students by email via the registrar's office, with one email per week for four weeks. The email will contain a link to a Callyope platform where the questionnaire can be completed. Students will create an account using their university email address as their username. If the student does not object, they will have to answer the first question of the questionnaire and then complete the full online questionnaire on the Callyope platform. The questionnaire will be available online on computers or smartphones for six weeks: from mid-October to the end of November. The questionnaire will be completed each year between mid-October and the end of November for the duration of the study or until the student completes their studies.

Duration of the inclusion period: 10 years Duration of participation for each participant: maximum 12 years Total duration of the study: 22 years

As the cohort progresses, longitudinal analyses may be conducted to study the evolution of various disorders over time, adjusting for known confounding factors. Following the initial analyses of this study, a new interventional study will be set up to identify students at risk and offer them appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Students who have been enrolled in first year of health studies at the University of Orléans
* Aged 18 or over

Exclusion Criteria:

* Does not speak French
* Person under legal guardianship
* Person deprived of liberty
* Person under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All students who were enrolled in their first year of health studies at the University of Orléans
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2047-10-31 (Estimated); Study Completion 2047-10-31 (Estimated)

PRIMARY OUTCOMES:
Measure Major Depressive Disorder prevalence | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  Measure of the 12-month Major Depressive Disorder prevalence by the Composite International Diagnostic Interview Short-Form (CIDI-SF).

SECONDARY OUTCOMES:
Measure prevalence of psychiatric disorders | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  Measure the annual prevalence of psychiatric disorders other than depression (anxiety, burnout, eating disorders, alcohol and cannabis addiction, childhood trauma) among medical students by comparing them to students who completed their first year but did not enter the medical.
  Anxiety will be assessed using the GAD7; eating disorders by the SCOFF, alcohol addiction by the AUDIT, cannabis addiction by the CUDIT, burnout by the MBI-SS (student version for pre-clinical students) or the MBI-HSS (caregiver version for externs and residents), and childhood trauma by the ACE.
Identify risk and protective factors for psychiatric disorders | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  Identify risk and protective factors for psychiatric disorders other than depression (anxiety, burnout, eating disorders, alcohol and cannabis addiction) among medical students by comparing them to students who completed their first year but did not enter the medical program.
  Anxiety will be assessed using the GAD7; eating disorders by the SCOFF, alcohol addiction by the AUDIT, cannabis addiction by the CUDIT, burnout by the MBI-SS (student version for pre-clinical students) or the MBI-HSS (caregiver version for externs and residents), and childhood trauma by the ACE.
Measure Major Depressive Disorder prevalence by year | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  Measure the prevalence of major depressive disorder each year among medical students by comparing them to students who have completed their first year but have not entered the medical program. Major Depressive Disorder prevalence will be measure by the Composite International Diagnostic Interview Short-Form (CIDI-SF).
Measure the prevalence of healthcare use and non-use | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  Measure the prevalence of healthcare use and non-use among medical students each year by comparing them to students who completed their first year but did not enter the medical program. Healthcare use will be assessed using questions from the WHO quality of life questionnaire, the Observatoire de la Vie Etudiants questionnaires, and the Mental Ill-ness : Clinicians' Attitudes (MICA).
Identify risk factors for non-use of healthcare | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  Identify risk factors for non-use of healthcare among medical students by comparing them to students who completed their first year but did not enter the medical program. Healthcare use will be assessed using questions from the WHO quality of life questionnaire, the Observatoire de la Vie Etudiants questionnaires, and the Mental Ill-ness : Clinicians' Attitudes (MICA).
Assess the stigma associated with psychiatric disorders | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  Assess the stigma associated with psychiatric disorders or the discipline of psychiatry among medical students by comparing them to students who completed their first year but did not enter the medical program. Stigma will be assessed using questions from the WHO quality of life questionnaire, the Observatoire de la Vie Etudiants questionnaires, and the Mental Ill-ness : Clinicians' Attitudes (MICA).
  Assessment of childhood trauma using the Adverse Childhood Experiences scale.
Factors of financial and social insecurity | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  Study the factors of financial and social insecurity (several variables) among medical students by comparing them to students who completed their first year but did not enter the medical program. Financial and social insecurity will be assessed using questions from the WHO quality of life questionnaire, the Observatoire de la Vie Etudiants questionnaires, and the Mental Ill-ness : Clinicians' Attitudes (MICA). Loneliness will be assessed using the UCLA loneliness
Assessment of educational support | Students fulfil the questionnaire on line once a year from enrollment until students complete their studies.
  For postgraduate students, assess their feelings about educational support.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmina MALLET, MD-PhD, Principal Investigator — CHOrléans
Locations (1):
- Centre Hospitalier Universitaire d'Orléans, Orléans, Loiret, France

REFERENCES:
- [Background] Husky MM, Leon C, du Roscoat E, Vasiliadis HM. Prevalence of suicidal thoughts and behaviors among young adults between 2000 and 2021: Results from six national representative surveys in France. Psychiatry Res. 2024 Mar;333:115763. doi: 10.1016/j.psychres.2024.115763. Epub 2024 Feb 1. PMID 38325160
- [Background] Frajerman A, Chevance A, Chaumette B, Morvan Y. Prevalence and factors associated with depression and suicidal ideation among French students in 2016: A national study. Psychiatry Res. 2023 Aug;326:115263. doi: 10.1016/j.psychres.2023.115263. Epub 2023 May 30. PMID 37295352
- [Background] Frajerman A, Rolland F, Hadouiri N, Haas-Jordache A, Gouy E, Mathieu L, Goulard A, Leon C, Morvan Y. Depression and suicidal thoughts in medical students and the general population: A comparison from 2 national studies. Gen Hosp Psychiatry. 2024 Sep-Oct;90:204-205. doi: 10.1016/j.genhosppsych.2024.07.002. Epub 2024 Jul 4. No abstract available. PMID 38997936
- [Background] Rolland F, Hadouiri N, Haas-Jordache A, Gouy E, Mathieu L, Goulard A, Morvan Y, Frajerman A. Mental health and working conditions among French medical students: A nationwide study. J Affect Disord. 2022 Jun 1;306:124-130. doi: 10.1016/j.jad.2022.03.001. Epub 2022 Mar 8. PMID 35276314
- [Background] Vergeron L, Morvan Y, Hadouiri N, Haas-Jordache A, Gouy E, Mathieu L, Goulard A, Rolland F, Frajerman A. Use of service and treatment adequacy in medical students and residents suffering from depression in France: A nationwide study. Psychiatry Res. 2024 Sep;339:115975. doi: 10.1016/j.psychres.2024.115975. Epub 2024 May 31. PMID 38875916
- [Background] Frajerman A. [Which interventions improve the well-being of medical students? A review of the literature]. Encephale. 2020 Feb;46(1):55-64. doi: 10.1016/j.encep.2019.09.004. Epub 2019 Nov 22. French. PMID 31767254
- [Background] Gosling CJ, Colle R, Cartigny A, Jollant F, Corruble E, Frajerman A. Measuring loneliness: a head-to-head psychometric comparison of the 3- and 20-item UCLA Loneliness Scales. Psychol Med. 2024 Oct 31;54(14):1-7. doi: 10.1017/S0033291724002083. Online ahead of print. PMID 39479755
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Garcia FD, Grigioni S, Chelali S, Meyrignac G, Thibaut F, Dechelotte P. Validation of the French version of SCOFF questionnaire for screening of eating disorders among adults. World J Biol Psychiatry. 2010 Oct;11(7):888-93. doi: 10.3109/15622975.2010.483251. PMID 20509759
- [Background] Gache P, Michaud P, Landry U, Accietto C, Arfaoui S, Wenger O, Daeppen JB. The Alcohol Use Disorders Identification Test (AUDIT) as a screening tool for excessive drinking in primary care: reliability and validity of a French version. Alcohol Clin Exp Res. 2005 Nov;29(11):2001-7. doi: 10.1097/01.alc.0000187034.58955.64. PMID 16340457
- [Background] Luquiens A, Berger-Viergat A, Larrieu A, Artigaud L, Fener C, Adamson S, Laprevote V, Rolland B. Validation of the French version of the Cannabis Use Disorder Identification Test-Revised and comparison with the Cannabis Abuse Screening Test for screening cannabis use disorder in a psychiatric sample. Drug Alcohol Rev. 2021 Nov;40(7):1334-1339. doi: 10.1111/dar.13298. Epub 2021 Apr 14. PMID 33855757
- [Background] Simon N, Verdoux H. [Impact of education program and clinical posting in psychiatry on medical students' stigmatizing attitudes towards psychiatry and psychiatric disorders]. Encephale. 2018 Sep;44(4):329-336. doi: 10.1016/j.encep.2017.05.003. Epub 2017 Jun 9. French. PMID 28606624